CLINICAL TRIAL: NCT06865261
Title: Effects of L-arginine and Liposomal Vitamin C Supplementation on Physical Performance and Endothelial Function in Elderly With Sarcopenia
Brief Title: Effects of L-ARGinine and Liposomal Vitamin C Supplementation On Physical Performance
Acronym: ARGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 6417
Record Dates: First submitted 2024-05-29; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-05

CONDITIONS: Sarcopenia
Keywords: aging; muscle wasting; physical function; handgrip; nitric oxide
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): the intervention group will receive twice-daily an oral supplementation with a combination of L-arginine 1.66 g plus liposomal Vitamin C 500 mg for 8 weeks
  Interventions: Dietary Supplement: Bioarginina C
- Control (Placebo Comparator): Control group will receive placebo twice a day for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bioarginina C — Bioarginine®C oral vials is a dietary supplement based on L-arginine and liposomal Vitamin C that is useful for making an integrative share of L-arginine and Vitamin C. Liposomal Vitamin C is a particular type of Vitamin C produced through an innovative technology that optimizes and amplifies its absorption.
  Arms: Experimental Group
Dietary Supplement: Placebo — Vials containing placebo were made to be indistinguishable in appearance from active treatment
  Arms: Control

SUMMARY:
In older age, reduced mobility is associated with an increased risk of reduced quality of life, disability, institutionalisation, and death, as well as increased healthcare expenditures. Sarcopenia is a condition characterised by a reduction in muscle mass and strength and/or function. It is associated with several adverse outcomes, such as falls, increased risk of infection, disability, institutionalisation, and death. Currently, no pharmacological treatments are available to combat sarcopenia. The management of sarcopenia relies on the adoption of an active lifestyle, comprising resistance exercise, which may be supported by an adequate intake of protein with the diet. Recently, treatment with L-arginine and liposomal vitamin C has been shown to significantly reduce fatigue, and improve physical performance and endothelial reactivity in adult patients with Long COVID. Long COVID may be considered a model of accelerated ageing, as it recapitulates several age-associated biological processes, including chronic inflammation, oxidative stress, endothelial dysfunction and malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* probable sarcopenia defined according to EWGSOP2 criteria

Exclusion Criteria:

* Inability or unwillingness to provide informed consent;
* NH residents;
* schizophrenia or other psychotic disorders, bipolar syndrome;
* consumption of more than 14 alcoholic beverages per week;
* reduced cognitive performance (Mini-Mental State Examination score <26);
* severe arthrosis;
* malignancies requiring treatment in the previous 3 years;
* lung disease requiring chronic corticosteroid therapy or oxygen therapy;
* severe cardiovascular disease;
* Parkinson's disease or other developmental neurological disorders;
* renal failure undergoing dialysis treatment;
* chest pain, severe dyspnea or conditions that may pose safety concerns when performing the 6-minute test or chair test;
* other medical, psychiatric or behavioral factors that, in the judgment of the researcher, may interfere with participation in the study;
* other illnesses related to an estimated life expectancy of less than 12 months.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
6MWT | 2 months
  Change from baseline to day 56 in the distance walked on the 6 min walk test

SECONDARY OUTCOMES:
HG | 2 months
  Change from baseline to day 56 in handgrip strength
CST | 2 months
  Change from baseline to day 56 in time to complete 5-repetition chair stand test
FMD | 2 months
  Change from baseline to day 56 in flow mediated dilation valuesbetween treatment and control group

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Tosato, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy